CLINICAL TRIAL: NCT04527302
Title: A Randomized Clinical Trial of Transcranial Direct Current Stimulation (tDCS) Concurrent With Exposure-based Cognitive-Behavioral Therapy (CBT) for Obsessive-Compulsive Disorder (OCD)
Brief Title: Efficacy of Augmentation of Cognitive Behavioral Therapy With Transcranial Direct Current Stimulation for Obsessive-Compulsive Disorder (OCD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-008
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: transcranial direct current stimulation; cognitive-behavioral therapy; Exposure and Response /Ritual Prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS+exposure based CBT (Active Comparator): The exposure and response prevention (ERP) treatment concurrently with an anode transcranial direct current stimulation over the mPFC will be applied 8 times (tDCS+ERP, 8sessions) in the whole treatment.
  Interventions: Combination Product: ERP combined with high-definition active tDCS
- sham tDCS +exposure based CBT (Sham Comparator): the exposure and response prevention (ERP) treatment concurrently with an sham transcranial direct current stimulation over the mPFC will be applied 8 times (sham tDCS+ERP, 8 sessions) in the whole treatment.
  Interventions: Combination Product: ERP combined with sham tDCS

INTERVENTIONS:
Combination Product: ERP combined with high-definition active tDCS — The active tDCS +ERP referred to a period of tDCS applied in the first 20 minutes of the ERP treatment (the tDCS device was activated when ERP began and deactivated automatically while ERP continued). The total treatment phase lasted eight weeks and included ten sessions with experienced psychotherapists following a specific manual for the tDCS+ERP treatment.
  The tDCS device will deliver a direct current of 1.5mA during 20 minutes. Anode electrode will be localized in front of the mPFC on the FpZ point according to the EEG international reference. Four cathode electrodes will be placed around (i.e. AF7, AF8, F3, F4).
  Arms: active tDCS+exposure based CBT
Combination Product: ERP combined with sham tDCS — Patients will get the same CBT setting as the active tDCS group and they were applied the sham tDCS cocurrently with ERP. The sham tDCS device is the same as the active comparator's except that the sham tDCS will only deliver a current stimulation for the first and last 15 seconds in order to produce somatic sensation in patients similar to that induced by the active tDCS.
  Arms: sham tDCS +exposure based CBT

SUMMARY:
This study aims to evaluate the feasibility and clinical outcome of the Exposure-based Cognitive-Behavioral Therapy (CBT) concurrent with Transcranial Direct Current Stimulation (tDCS) in treating obsessive-compulsive disorder (OCD) patients, and explores the potential neural mechanisms of treatment effect by magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
The current study aims to evaluate feasibility and clinical outcome of exposure-based CBT（ERP）combined with tDCS over the prefrontal cortex (mPFC) in treatment of OCD patients. 60 OCD patients whose symptom were mainly associated with "contamination/clean" will be randomized into two groups (i.e. ERP+active tDCS or ERP+sham tDCS stimulation). Over a two-month period, all patients are received 10 sessions of individual CBT, including 8 sessions of concurrent tDCS with ERP (tDCS+ERP). Three independent evaluators will rate the severity of patients' obsessive-compulsive symptoms using Y-BOCS at four assessment points: baseline (prior to the treatment), after the first (session 2#), fourth (session 5#), and eighth treatment of tDCS+ERP (session 10#). The patients will also receive MRI scan and EEG.

The current study aims to explore whether the administration of online tDCS together with ERP (tDCS+ERP) will improve the efficacy of ERP and tries to provide some early evidience that reveal potential neural mechanisms of the treatment.

ELIGIBILITY:
We recruited outpatient adults with OCD confirmed by the Mini-International Neuropsychiatric Interview (MINI). The following inclusion and exclusion criteria were also applied:

Inclusion Criteria:

(1) 18-50 years old, with at least 9 years of education, (2) Y-BOCS score ≥16, (3) no history of serious medical, neurological illness or other psychotic disorders other than OCD (anxiety or mild to moderate depression secondary to OCD was not exclusionary), (4) medication-free or had received stable medication for at least 2 months before entering the study and continued the same medication throughout the study (5) no previous exposure to ERP or tDCS.

Exclusion Criteria:

* history of serious medical, neurological illness or other psychotic disorders other than OCD
* The inability to receive tDCS because of metallic implants, or history of seizures，or history of head injury, or history of neurosurgery.
* Participants who have received ECT, rTMS, tDCS and CBT in the past.
* Participants with claustrophobic, heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.
* serious suicide risk

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was represented by the percent reduction of Y-BOCS scores | baseline，2 weeks，4 weeks to 8 weeks (pre-treatment, after Session 2, 5, 10)
  We defined the tDCS+ERP treatment response as the percent reduction of Y-BOCS scores greater than or equal to 35%.

SECONDARY OUTCOMES:
Change in Obsessive Compulsive Inventory-Revised(OCI-R) | baseline，2 weeks，4 weeks to 8 weeks(pre-treatment, after Session 2, 5, 10)
  It is an inventory of OCD symptoms with 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Change in Beck Depression Inventory(BDI) | baseline，2 weeks，4 weeks to 8 weeks(pre-treatment, after Session 2, 5, 10)
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in Beck Anxiety Inventory (BAI) | baseline，2 weeks，4 weeks to 8 weeks(pre-treatment, after Session 2, 5, 10)
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Change in Perceived Stress Scale(PSS) | baseline，2 weeks，4 weeks to 8 weeks(pre-treatment, after Session 2, 5, 10)
  It is a 10-item, 5-point Likert scale(0 to 4) to measure the degree to which situations in one's life are appraised as stressful.The total score ranges from 0 to 40, with lower total scores representing a better outcome.
Change in Pittsburgh sleep quality index(PSQI) | baseline，2 weeks，4 weeks to 8 weeks(pre-treatment, after Session 2, 5, 10)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Change in Side-effect questionnaire | 2 weeks，4 weeks to 8 weeks(after Session 2, 5, 10)
  It consists of 10-item and uses 0 to 3 severity scale to rate the intensity of side effects. Total scores range from 0 to 30, with higher scores indicating more severe side-effect. It also assesses the relation between side-effect and the effects of tDCS using 0 to 4 scale. Total scores range from 0 to 40, with higher score indicating the greater relation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China